CLINICAL TRIAL: NCT04378660
Title: Artificial Intelligence Validation Trial for Polyp Detection: Pilot Study
Brief Title: Artificial Intelligence (AI) Validation Study for Polyp Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Nuovo Regina Margherita Hospital, Rome, Italy (Unknown); Universitäts Medizin, Mainz, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: s59405
Record Dates: First submitted 2020-04-20; First posted 2020-05-07 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-04

CONDITIONS: Polyp of Colon
Keywords: Colonic polyp; Artificial intelligence; Second observer
MeSH Terms: conditions — Colonic Polyps | interventions — Artificial Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Colonoscopy with AI
  Interventions: Diagnostic Test: Artificial intelligence for polyp detection

INTERVENTIONS:
Diagnostic Test: Artificial intelligence for polyp detection — Colonoscopy enriched with artificial intelligence tool developed for polyp detection, implemented as a second observer

SUMMARY:
Interventional prospective multicenter study: Polyp detection by an automated endoscopic tool as second observer during routine diagnostic colonoscopy

DETAILED DESCRIPTION:
This is an investigator-initiated multicentre non-randomized prospective interventional trial to validate the performance of a novel state-of-the-art computer-aided diagnostic (CAD) tool in polyp detection implemented as second observer during routine diagnostic colonoscopy and to evaluate its feasibility in daily endoscopy. Patients referred for a screening surveillance or therapeutic colonoscopy will undergo a colonoscopy performed by an endoscopist with moderate to high adenoma detection rate (ADR > 20% and < 50%) while a second observer will follow the procedure on a bedside AI-tool to count the number of detections made by the AI system and categorize the results into positive or negative results as follows (1) true positive, (2) false negative, (3) other positive and (4) obvious false positive. When a doubtful detection is made by the AI-system, the second observer will ask to re-evaluate the indicated region. When the detection is clear, the endoscopist and second observer do not communicate. The entire procedure is recorded.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* Diagnostic or screening colonoscopy
* Therapeutic colonoscopy

Exclusion Criteria:

* Inability to give informed consent by the patient or legal representative
* < 18 years old
* Any contraindication for colonoscopy or biopsies of the colon
* Uncontrolled coagulopathy
* Confirmed diagnosis of inflammatory bowel disease
* Short bowel or ileostomy
* Pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-04-18 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of the novel AI system compared to endoscopic diagnosis as gold standard | 4 months
  Determination of the diagnostic accuracy of the novel AI system as second observer

SECONDARY OUTCOMES:
Endoscopist's polyp miss rate as number of extra AI detections | 4 months
  Determination of the AI system's precision and extra value as second observer

CONTACTS AND LOCATIONS:
Overall Officials: Raf Bisschops, Principal Investigator — UZ Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No
We don't share any patient information with other researchers, nor when it's anonymized

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-30): https://cdn.clinicaltrials.gov/large-docs/60/NCT04378660/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT04378660/ICF_001.pdf